CLINICAL TRIAL: NCT01313104
Title: Pilot Project for Anal Dysplasia Screening in Women With Cervical or Vulvar Dysplasia
Brief Title: Colposcopy and High Resolution Anoscopy in Screening For Anal Dysplasia in Patients With Cervical, Vaginal, or Vulvar Dysplasia or Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NU 10G02; NCI-2011-00112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00039225 (Other: Northwestern University IRB)
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 1; Cervical Intraepithelial Neoplasia Grade 2; Cervical Intraepithelial Neoplasia Grade 3; Recurrent Cervical Cancer; Recurrent Vaginal Cancer; Recurrent Vulvar Cancer; Stage 0 Cervical Cancer; Stage 0 Vaginal Cancer; Stage 0 Vulvar Cancer; Stage I Vaginal Cancer; Stage I Vulvar Cancer; Stage IA Cervical Cancer; Stage IB Cervical Cancer; Stage II Vaginal Cancer; Stage II Vulvar Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage III Vaginal Cancer; Stage III Vulvar Cancer; Stage IV Vulvar Cancer; Stage IVA Cervical Cancer; Stage IVA Vaginal Cancer; Stage IVB Cervical Cancer; Stage IVB Vaginal Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Colposcopy; Vaginal Smears; High-Throughput Screening Assays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening (Experimental): See Detailed Description
  Interventions: Procedure: colposcopy; Other: cervical Papanicolaou test; Procedure: screening method

INTERVENTIONS:
Procedure: colposcopy — Undergo colposcopy
Other: cervical Papanicolaou test — Undergo cervical Pap smear
  Other Names: cervical Pap test
Procedure: screening method — Undergo anal Pap smear
Procedure: screening method — Undergo high resolution anoscopy

SUMMARY:
This clinical trial studies colposcopy and high resolution anoscopy in screening for anal dysplasia in patients with cervical, vaginal, or vulvar dysplasia or cancer. Screening may help doctors find cancer cells early and plan better treatment for cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the risk of anal dysplasia in women with cervical or vulvar dysplasia.

OUTLINE:

Patients undergo colposcopy and cervical Papanicolaou test with Human papillomavirus (HPV) test followed by anal Papanicolaou test and high resolution anoscopy. Patients with dysplastic anal lesions undergo repeat anoscopy at 3, 9, 15, and 24 months. Patients with normal anoscopy are followed up at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of cervical, vaginal or vulvar intraepithelial neoplasia or cancer are included
* Individuals treated with prior radiation therapy and/or chemotherapy are allowed
* Women with high-grade dysplasia (carcinoma in situ) are eligible, regardless of their dysplasia free interval
* HIV-positive (Human Immunodeficiency Virus) and HIV-negative women will be enrolled; HIV testing will not be performed as part of the study

Exclusion Criteria:

* Women who are not able to consent are excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Risk of anal dysplasia in women with cervical or vulvar dysplasia | Over 2 years
HPV (Human Papillomavirus) status | Over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amy Halverson, Principal Investigator — Northwestern University